CLINICAL TRIAL: NCT03455049
Title: The Effect of Andrographis Paniculata to GLP-1, Fasting Insulin, Insulin 2-h Post OGTT, and HOMA-IR in Normal and Prediabetes Subject
Brief Title: The Effect of Andrographis Paniculata to GLP-1, Fasting Insulin, Insulin 2-h Post OGTT, and HOMA-IR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr Tri Juli Edi Tarigan, SpPD-KEMD, MD, Endocrinologist, Indonesia University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaU-02
Record Dates: First submitted 2018-01-17; First posted 2018-03-06 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Increased Insulin
MeSH Terms: conditions — Hyperinsulinism

STUDY DESIGN:
Intervention Model Description: Clinical Trials with Randomization, Double Blind, Crossover
Who Masked: Participant, Investigator
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Normal subject experimental (Experimental): Participants get Andrographis Paniculata Extract 550 mg, two capsules, twice a day, for 14 days.
  Interventions: Other: Andrographis Paniculata Ext
- Normal subject placebo (Placebo Comparator): Participants get placebo consist of Lactose 98%, Mg 2%, two capsules, twice a day, for 14 days.
  Interventions: Other: Andrographis Paniculata Ext
- Prediabetes subject experimental (Experimental): Participants get Andrographis Paniculata Extract 550 mg, two capsules, twice a day, for 14 days.
  Interventions: Other: Andrographis Paniculata Ext
- Prediabetes subject placebo (Placebo Comparator): Participants get placebo consist of Lactose 98%, Mg 2%, two capsules, twice a day, for 14 days.
  Interventions: Other: Andrographis Paniculata Ext

INTERVENTIONS:
Other: Andrographis Paniculata Ext — Give the Androgaphis paniculata in prediabetes and normal subject for 14 days.

SUMMARY:
Prevalence of type 2 diabetes have been increased, but medications had not been well, so that needed new alternatives. A new approach used in management of type 2 diabetes is incretin based therapy. Incretin hormone, glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotrophic peptide (GIP), had producted in intestine due to carbohydrate intralumen. After had secreted, GLP-1 had degradated by DPP-4 enzyme till number and effect had been decreased. Decreasing of GLP-1 effect as main defect in type 2 diabetes.

Andrographis paniculata (A. paniculata) as traditional treatment had known since years ago to have hypoglycemia effect. Extract of A. paniculata consists of andrographolid and flavonoid. Based on study of Wooten et al that flavonoid has hydroxyl to stimulate insulin's production through modulated GLP-1 receptor (GLP-1 receptor ligand). So the investigators need to study about The Effect of A. paniculata Extract to GLP-1, Fasting Plasma Insulin, Insulin concentrations measured during a standardized 2-h OGTT, and HOMA-IR.

DETAILED DESCRIPTION:
Blood's participants will be examined fasting plasma insulin and glycated albumin (from fasting blood) and insulin measured during a standardized 2-h OGTT, DPP-4 enzyme, and GLP-1 (from standardized 2-h OGTT blood). Then, complete urinalysis test. Participants will be randomized to be two groups are group have been intervenced by capsules of A. paniculata or group placebo. Each group will be explained about procedure to consume capsules A. paniculata or placebo for 14 days, storage procedures, and the way to contact the investigators if adverse event happened. The investigators will contact participants to remember the schedule to consume capsules A. paniculata, ask whether the side effects or not, and ask the result of self monitoring blood glucose every three days by glucose meter have been given.

Before day 12th, participants will be contacted to come in visit 2nd. In visit 2nd (day 15th) will be done anamneses, assessment of compliance, reporting adverse event and side effect, physical examination, fasting plasma glucose test, fasting insulin, HOMA-IR, GA and complete urinalysis. Then, will be done standardized 2-h OGTT. Two hours later, it will be done plasma glucose level, insulin, DPP-4 enzyme, and GLP-1. Participants will be explained that they will not receive capsules of A. paniculata for 7 days (day 15th till 21th). This is called wash out.

Participants will be explained about procedures to consume capsule of A. paniculata or placebo in day 22th till 35th. Before day 32th, participants will be contacted to come in visit 3rd (day 36th). In visit 3rd, will be done anamneses, assessment of compliance, reporting adverse event and side effect, physical examination, fasting plasma glucose test, fasting insulin, HOMA-IR, GA and complete urinalysis. Then, will be done standardized 2-h OGTT. Two hours later, it will be done plasma glucose level, insulin, DPP-4 enzyme, and GLP-1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 year old until 60 year old
2. Normal glucose tolerance subject or prediabetes
3. The kidney function (creatinine) and liver function (SGPT) in range normal
4. Subject has signed agreement (informed consent)

Exclusion Criteria:

1. Pregnant
2. Feeding baby
3. Subject has comorbide or chronic disease uncontrolled
4. Subject has cancer
5. Subject consume medication influenced blood glucose such as steroid an suplement
6. Insulin dependent diabetes

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-02 (Actual)

PRIMARY OUTCOMES:
GLP-1 | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes incretin effect

SECONDARY OUTCOMES:
Fasting Insulin | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes beta-cell secretion
2h-OGTT Insulin | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes beta-cell secretion after 2h-OGTT
HOMA-IR | A measure assesing change from baseline GLP-1 at 14 days.
  Index of insulin resistance
Fasting plasma glucose level | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes beta-cell function
2h-OGTT plasma glucose level | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes beta-cell function after 2h-OGTT
Dypeptidil Peptidase 4 (DPP-4) Enzyme | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes degradation of GLP-1 in Ileum
Glycated Albumin | A measure assesing change from baseline GLP-1 at 14 days.
  Index analyzes plasma glucose during 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tri Juli Edi Tarigan, MD, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wedick NM, Pan A, Cassidy A, Rimm EB, Sampson L, Rosner B, Willett W, Hu FB, Sun Q, van Dam RM. Dietary flavonoid intakes and risk of type 2 diabetes in US men and women. Am J Clin Nutr. 2012 Apr;95(4):925-33. doi: 10.3945/ajcn.111.028894. Epub 2012 Feb 22. PMID 22357723
- [Derived] Tarigan TJE, Purwaningsih EH, Yusra, Abdullah M, Nafrialdi, Prihartono J, Saraswati MR, Subekti I. Effects of Sambiloto (Andrographis paniculata) on GLP-1 and DPP-4 Concentrations between Normal and Prediabetic Subjects: A Crossover Study. Evid Based Complement Alternat Med. 2022 Jan 15;2022:1535703. doi: 10.1155/2022/1535703. eCollection 2022. PMID 35075363